CLINICAL TRIAL: NCT05704660
Title: Retraining the Automatic Reaction to Physical Activity and Sedentary Stimuli in Adults 60 Years of Age or Older
Brief Title: Automatic Reaction to Physical Activity and Sedentary Stimuli in Aging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Matthieu Boisgontier, Principal Investigator, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H-09-22-8453
Record Dates: First submitted 2023-01-10; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Aging
Keywords: Attentional Bias; Exercise; Sedentary Behavior
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and research assistant will be blinded to the groups' allocation. The participant blinding success will be appraised by asking them to guess in what group there were at the trial termination. Besides, the research assistant blinding success will be appraised via detecting the group allocation (Experimental vs. Control) by research assistant at the end of data collection phase. The randomization will be generated on a computer and an independent coworker will carry out the randomization. The participant's identification number will be used to determine the sequence of randomization. Participants will be randomized in a 1:1 ratio between the intervention and active control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjusted and modified Cognitive-Biased Modification Task (Experimental): The intervention is based on a Go/No-Go task.
  Interventions: Behavioral: Adjusted Cognitive-biased modification task
- Normal Cognitve-Biased modification Task (Placebo Comparator): The Sham-intervention is based on a Go/No-Go task.
  Interventions: Behavioral: Cognitive-biased modification task

INTERVENTIONS:
Behavioral: Adjusted Cognitive-biased modification task — The intervention of the proposed project is based on a go/no-go task in which older adults need to quickly decide whether or not they should react to the stimulus. A rectangle containing an image, or a word will be presented on a screen. In the intervention group, older adults will be instructed to restrain their actions when the rectangle is tilted to the right and to react by pressing a key on the keyboard when the rectangle is tilted to the left, irrespective of the content of the rectangle (because the training is meant to be implicit). In order to train inhibitory processes counteracting the automatic attraction to sedentary behavior, 90% of the rectangles tilted to the right (counterbalanced across participants) will contain a picture or a word related to sedentary behavior. To foster the automatic attraction toward physical activity, 90% of the rectangles tilted to the left will contain a picture or a word related to physical activity.
  Arms: Adjusted and modified Cognitive-Biased Modification Task
Behavioral: Cognitive-biased modification task — In the comparison group, instructions will be identical, but the percentage of physical activity and sedentary stimuli will be equal in each tilt condition (i.e., 50% sedentary stimuli and 50% physical activity stimuli in both right- and left-tilted rectangles)
  Arms: Normal Cognitve-Biased modification Task

SUMMARY:
Most individuals are aware of the benefits to health of regular physical activity and have good intentions to exercise. Yet, 1.4 billion people worldwide are inactive, which suggests that turning intention into action can be challenging. Recent findings show that the intention-action gap could be explained by negative automatic reactions (which is a component of dual-task theory) to stimuli associated with physical activity. This gap is particularly concerning in older adults, who are more likely to spontaneously associate physical activity with fear, pain, or discomfort. To promote physical activity, the current project proposes to train older adults to suppress their automatic attraction toward sedentary stimuli and to respond positively to physical-activity stimuli. This evidence-based and low-cost intervention aims to improve physical functioning and quality of life for these population. The results will inform public-health policies and improve clinical interventions that aim to counteract a global health problem: the pandemic of physical inactivity.

DETAILED DESCRIPTION:
Physical activity is one of the top contributors to health, reducing rates of cardiovascular disease, cancer, hypertension, diabetes, obesity, and depression. This wide spectrum of benefits is particularly important for older adults, who often suffer structural and functional deterioration in several physiological systems. Physical activity can reduce and delay the impact of this age-related deterioration in health and functional independence. Current interventions to enhance physical activity in older adults rely mainly on reflective processes by providing rational information about the health benefits of a physically active lifestyle. While these interventions successfully increase intention, their effect on actual behavior is weak. That is, most individuals are now aware of the positive effects of regular physical activity and have the intention to exercise. However, this intention is not sufficient and exercise plans are often not executed. This gap between intention and action is a challenge that health professionals need to address to counteract the pandemic of physical inactivity. Recent findings suggest that this inability to turn the intention into action is explained by negative automatic reactions to stimuli associated with physical activity. These automatic reactions could be particularly strong in older adults, who are more likely to associate physical activity with fear, pain, or discomfort. This study aims to test the effect of an intervention that targets the automatic processes underlying physical inactivity in older adults. The intervention is expected to reduce physical inactivity during the intervention and at follow-up, thereby improving physical functioning and quality of life.

ELIGIBILITY:
Inclusion Criteria:

- 60 years of age or older and able to understand instructions in English.

Exclusion Criteria:

* Diagnosed psychiatric disorders or neurological condition (e.g., stork, Parkinson's disease, Alzheimer's disease, dementia)
* Unable to carry out the training program
* Unable to understand the protocol
* Motor deficit preventing physical activity without external help
* Physical health status preventing physical activity
* Alcohol or substance dependence.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Physical activity Tracker | "7 days", at least "7 hours" per day (not to used it during shower or when they sleep at night).
  Assessing the number of step.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire (Short Form) | Before and after intervention ("10 minutes" to fill out)
  The usual level of moderate-to-vigorous physical activity in minutes per week will be assessed.
Six-Minute Walk Test | Before and after intervention ("6 minutes" to carry out)
  Total distance walked in "6 minutes" will be documented. The outcome is the distance walked during the "6 minutes".
Hand grip strength | Before and after intervention ( "One minute" to carry out)
  The grip strength will be evaluated using a dynamometer. The higher the value obtained by the participant, the stronger the grip.
World Health Organization Quality of Life (BREF) | Before and after intervention ( "20 minutes" to carry out)
  Assessing quality of life over four domains. Scores for each domain can range from zero to 100, with higher scores indicating better quality of life.
Approach-avoidance task | Before and after intervention, and at the beginning of each intervention session ("30 minutes" to carry out)
  To measure automatic approach and avoidance tendencies toward physical activity and sedentary behaviors. Faster and the more accurate reaction toward a stimuli (e.g., physical activity) indicates a stronger tendency to approach that specific stimuli.
Explicit Affective Attitude Toward Physical Activity | Before and after intervention ("2-5 minute" to carry out)
  Mean of two items based on two "7-point" scales (unpleasant-pleasant; unenjoyable-enjoyable). A higher score indicates more positive attitudes toward physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu P Boisgontier, PhD, Principal Investigator — University of Ottawa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guthold R, Stevens GA, Riley LM, Bull FC. Worldwide trends in insufficient physical activity from 2001 to 2016: a pooled analysis of 358 population-based surveys with 1.9 million participants. Lancet Glob Health. 2018 Oct;6(10):e1077-e1086. doi: 10.1016/S2214-109X(18)30357-7. Epub 2018 Sep 4. PMID 30193830
- [Background] Kohl HW 3rd, Craig CL, Lambert EV, Inoue S, Alkandari JR, Leetongin G, Kahlmeier S; Lancet Physical Activity Series Working Group. The pandemic of physical inactivity: global action for public health. Lancet. 2012 Jul 21;380(9838):294-305. doi: 10.1016/S0140-6736(12)60898-8. PMID 22818941
- [Background] Cheval B, Boisgontier MP. The Theory of Effort Minimization in Physical Activity. Exerc Sport Sci Rev. 2021 Jul 1;49(3):168-178. doi: 10.1249/JES.0000000000000252. PMID 34112744
- [Background] Wiers RW, Eberl C, Rinck M, Becker ES, Lindenmeyer J. Retraining automatic action tendencies changes alcoholic patients' approach bias for alcohol and improves treatment outcome. Psychol Sci. 2011 Apr;22(4):490-7. doi: 10.1177/0956797611400615. Epub 2011 Mar 9. PMID 21389338
- [Background] Wittekind CE, Feist A, Schneider BC, Moritz S, Fritzsche A. The approach-avoidance task as an online intervention in cigarette smoking: a pilot study. J Behav Ther Exp Psychiatry. 2015 Mar;46:115-20. doi: 10.1016/j.jbtep.2014.08.006. Epub 2014 Sep 16. PMID 25306247
- [Background] Taylor CT, Amir N. Modifying automatic approach action tendencies in individuals with elevated social anxiety symptoms. Behav Res Ther. 2012 Sep;50(9):529-36. doi: 10.1016/j.brat.2012.05.004. Epub 2012 May 23. PMID 22728645
- [Background] Aulbach MB, Knittle K, Haukkala A. Implicit process interventions in eating behaviour: a meta-analysis examining mediators and moderators. Health Psychol Rev. 2019 Jun;13(2):179-208. doi: 10.1080/17437199.2019.1571933. Epub 2019 Feb 6. PMID 30676235
- [Background] Cheval B, Radel R, Neva JL, Boyd LA, Swinnen SP, Sander D, Boisgontier MP. Behavioral and Neural Evidence of the Rewarding Value of Exercise Behaviors: A Systematic Review. Sports Med. 2018 Jun;48(6):1389-1404. doi: 10.1007/s40279-018-0898-0. PMID 29556981
- [Background] Cheval B, Tipura E, Burra N, Frossard J, Chanal J, Orsholits D, Radel R, Boisgontier MP. Avoiding sedentary behaviors requires more cortical resources than avoiding physical activity: An EEG study. Neuropsychologia. 2018 Oct;119:68-80. doi: 10.1016/j.neuropsychologia.2018.07.029. Epub 2018 Jul 26. PMID 30056055
- [Background] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Background] Haseler C, Crooke R, Haseler T. Promoting physical activity to patients. BMJ. 2019 Sep 17;366:l5230. doi: 10.1136/bmj.l5230. No abstract available. PMID 31530549
- [Background] Rhodes RE, Dickau L. Experimental evidence for the intention-behavior relationship in the physical activity domain: a meta-analysis. Health Psychol. 2012 Nov;31(6):724-7. doi: 10.1037/a0027290. Epub 2012 Mar 5. PMID 22390739
- [Background] Calitri R, Lowe R, Eves FF, Bennett P. Associations between visual attention, implicit and explicit attitude and behaviour for physical activity. Psychol Health. 2009 Nov;24(9):1105-23. doi: 10.1080/08870440802245306. PMID 20205048
- [Background] Conroy DE, Hyde AL, Doerksen SE, Ribeiro NF. Implicit attitudes and explicit motivation prospectively predict physical activity. Ann Behav Med. 2010 May;39(2):112-8. doi: 10.1007/s12160-010-9161-0. PMID 20140542
- [Background] Cheval B, Sarrazin P, Isoard-Gautheur S, Radel R, Friese M. Reflective and impulsive processes explain (in)effectiveness of messages promoting physical activity: a randomized controlled trial. Health Psychol. 2015 Jan;34(1):10-9. doi: 10.1037/hea0000102. Epub 2014 Aug 18. PMID 25133840

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/60/NCT05704660/Prot_SAP_ICF_000.pdf